CLINICAL TRIAL: NCT04880239
Title: REDUCE Trial - Reducing Prolapse Recurrence by Reducing the Genital Hiatus
Brief Title: REDUCE Trial- Reducing Prolapse Recurrence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: The Institute of Pelvic Medicine & Reconstructive Surgery, Allentown, Pennsylvania (Other); University of Kansas (Other)
Responsible Party: Principal Investigator, Julia Geynisman-Tan, Director of Research; Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00214588
Record Dates: First submitted 2021-04-14; First posted 2021-05-10 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Prolapse; Female
MeSH Terms: conditions — Prolapse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacralcolpopexy with posterior colpoperineorrhaphy (Active Comparator)
  Interventions: Procedure: Posterior colpoperineorrhaphy
- Sacralcolpopexy without posterior colpoperineorrhaphy (No Intervention)

INTERVENTIONS:
Procedure: Posterior colpoperineorrhaphy — Patients having a sacralcolpopexy will be randomized to ultra lightweight mesh (Coloplast Restorelle) with posterior colpoperineorrhaphy or the same procedure without the posterior colpoperineorrhaphy
  Arms: Sacralcolpopexy with posterior colpoperineorrhaphy

SUMMARY:
This study will examine whether surgeons should add a prophylactic posterior colpoperineorrhaphy to a mesh-augmented apical prolapse repair.

DETAILED DESCRIPTION:
The decision to perform a posterior colpoperineorrhaphy at the time of sacrocolpopexy is controversial. Based on cohort data, some surgeons advocate that sacrocolpopexy alone is effective at treating posterior vaginal wall prolapse and the addition of posterior colpoperineorrhaphy only increases the likelihood of pain with defecation and dyspareunia. Experts theorize that placement of posterior vaginal mesh down to the perineal body provides adequate posterior support and reduces genital hiatus size. Others argue that placement of mesh too low on the posterior vagina may be associated with increased mesh exposure and pain secondary to mesh stiffness. No randomized trials exist comparing prolapse outcomes using new, ultra-light polypropylene mesh with and without posterior colpoperineorrhaphy. The investigators hypothesize that there will be no difference in prolapse outcomes after sacrocolpopexy using Restorelle mesh with and without posterior colpoperineorrhaphy. However, patients with a posterior colpoperineorrhaphy will be more likely to report pain with defecation and dyspareunia. This will be the first multicenter randomized trial comparing outcomes of sacrocolpopexy with and without posterior colpoperineorrhaphy.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 18
* English or Spanish speaking
* Symptomatic prolapse (stage II or greater) undergoing minimally-invasive sacrocolpopexy with Restorelle ultra lightweight mesh
* Preoperative genital hiatus with valsalva/strain greater than or equal to 4cm

Exclusion Criteria:

* Patient has had prior prolapse surgery
* Patient has inflammatory bowel disease (Crohn's, Ulcerative Colitis)
* Baseline dyspareunia (patient reports that they have pain with vaginal intercourse when asked as a yes/no)
* Patients with a score of 7 or greater in any one muscle on the Meister Pelvic Floor Exam
* Patient planning a concomitant Burch procedure
* Pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-11-23 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Pelvic Organ Prolapse Quantification (POP-Q) System | 1 Year
  The POP-Q System will be used to compare the rate of prolapse recurrence at 1 year between women undergoing a sacrocolpopexy with Restorelle mesh with and without a concomitant posterior colpoperineorrhaphy.

SECONDARY OUTCOMES:
Defecatory Dysfunction | 1 Year
  To compare the rates of defecatory dysfunction using the Bristol Stool Scale (stool types measured from type 1-type 7) and the Colorectal-Anal Distress Inventory 8 (measured from 0-100 points).
Dyspareunia | 1 Year
  To compare the rates of dyspareunia between groups using the Female Sexual Function Index (measured from 2-36 points)
Surgical and Perioperative Events: Blood Loss | 2 Weeks
  To compare the estimated blood loss (in milliliters) between groups.
Surgical and Perioperative Events: Operative Time | Day of surgery
  To compare the operative time (in minutes as listed on the surgical case tracking) between groups.
Surgical and Perioperative Events: Postoperative Pain | 2 Weeks
  To compare postoperative pain scores using a visual analog scale (0-100 points) between groups.
Surgical and Perioperative Events: Pain Medication Use | 2 Weeks
  To compare narcotic pain medication use (in morphine equivalents consumed and reported by patients) between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Geynisman-Tan, M.D, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No